CLINICAL TRIAL: NCT05804318
Title: Daily Adaptive Stereotactic Body Radiation Therapy for Prostate Cancer With Urethral Sparing: A Prospective Trial Using an Individualized Approach to Reduce Urinary Toxicity
Brief Title: Daily Adaptive Radiation Therapy Using an Individualized Approach for Prostate Cancer
Acronym: ARTIA-Prostate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAR-2021-10
Record Dates: First submitted 2023-03-10; First posted 2023-04-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Adaptive SBRT with Urethral Sparing (Experimental): Daily adaptive stereotactic body radiation therapy delivering 40 Gy in 5 fractions to the prostate while delivery 35-36 Gy in 5 fractions to the urethra.
  Interventions: Device: Daily adaptive SBRT with urethral sparing

INTERVENTIONS:
Device: Daily adaptive SBRT with urethral sparing — The radiation plan for each daily fraction is adapted from the initial plan based on cone beam CT imaging acquired while the participant is laying on the treatment machine.

SUMMARY:
This trial is a prospective, single-arm, multi-center clinical trial designed to assess whether adaptive radiotherapy with urethral sparing for low to intermediate risk localized prostate cancer will translate into a decreased rate of patient reported acute urinary side effects, as measured by the patient reported EPIC-26 questionnaire, compared with the historically reported rate for non-adaptive, non-urethral sparing prostate SBRT.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has NCCN low or intermediate risk prostate cancer that is biopsy proven.
2. Prostate volume is ≤80cc as assessed by MRI prior to radiotherapy.
3. AUA/IPSS score is ≤ 15.
4. ECOG performance status is ≤2 (or Karnofsky score is ≥60%).
5. Patient has no PIRADS 4 or 5 lesion on prostate MRI contacting the urethra (determined at physician discretion).
6. Patient has the ability to complete required patient questionnaires.
7. Patient age ≥ 18 years (or greater than the local age of majority).
8. Patient has the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patient has baseline grade ≥3 GI or GU toxicity
2. Patient has had prior overlapping pelvic radiotherapy.
3. Patient has had prior transurethral resection of the prostate, prostate HIFU, or cryoablation.
4. Patient has node positive prostate cancer.
5. Patient has extracapsular extension (capsular abutment is permitted).
6. Patient has active inflammatory bowel disease or active collagen vascular disease.
7. Patient cannot undergo prostate MRI.
8. Patient cannot undergo prostate fiducial marker placement.
9. Patient has ongoing receipt of cytotoxic chemotherapy (androgen deprivation therapy is allowed).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Patient-reported acute urinary toxicity | 90 days after end of SBRT
  Minimum clinically important change (MCIC) status in patient-reported urinary QOL, as determined by the worst change reported by each subject in their EPIC-26 urinary domain scores.

SECONDARY OUTCOMES:
Freedom from biochemical recurrence | 5 years after end of SBRT
  Rate of biochemical recurrence free survival, as determined by the Phoenix definition (PSA level of 2 ng/ml or more higher than the lowest post-SBRT value)
Patient-reported quality of life issues related to prostate cancer. | Baseline; during treatment; 6 weeks, 3 months, 6 months, 12 months, 18 months, 2 years, 3 years, 4 years, and 5 years after end of SBRT
  Patient-reported quality of life changes during and after adaptive prostate SBRT treatment using the Expanded Prostate Cancer Index Composite Short Form (EPIC-26) questionnaire.
Patient-reported erectile dysfunction symptoms | Baseline; during treatment; 6 weeks, 3 months, 6 months, 12 months, 18 months, 2 years, 3 years, 4 years, and 5 years after end of SBRT
  Patient-reported erectile dysfunction symptoms before, during and after adaptive prostate SBRT treatment using the Sexual Health Inventory for Men (SHIM) questionnaire.
Patient-reported urinary symptoms | Baseline; during treatment; 6 weeks, 3 months, 6 months, 12 months, 18 months, 2 years, 3 years, 4 years, and 5 years after end of SBRT
  Patient-reported urinary symptoms before, during and after adaptive prostate SBRT treatment using the International Prostate Symptom Score (IPSS) questionnaire.
Patient-reported overall quality of life | Baseline; during treatment; 6 weeks, 3 months, 6 months, 12 months, 18 months, 2 years, 3 years, 4 years, and 5 years after end of SBRT
  Patient-reported overall quality of life before, during and after adaptive prostate SBRT treatment using the EQ-5D-5L questionnaire.
Physician-reported toxicities | During treatment; 6 weeks, 3 months, 6 months, 12 months, 18 months, 2 years, 3 years, 4 years, and 5 years after end of SBRT
  Physician-reported CTCAE v 5.0 adverse events
Alpha-blocker medication use | Baseline; during treatment; 6 weeks, 3 months, 6 months, 12 months, 18 months, 2 years, 3 years, 4 years, and 5 years after end of SBRT
  Change in use of alpha-blocker medications for urinary symptoms
Metastasis-free survival | 5 years after end of SBRT
  Metastasis-free survival
Prostate-cancer specific mortality | 5 years after end of SBRT
  Prostate-cancer specific mortality
Overall survival | 5 years after end of SBRT
  Overall survival
Workflow metrics of adaptive SBRT for prostate cancer | 2 weeks after start of SBRT
  Includes the time on table and frequency of using the adapted vs. non-adapted treatment plan for each fraction.
Target and OAR dosimetry | 2 weeks after start of SBRT
  Improvement in target coverage and/or reduction in dose to critical organs at risk in the adapted plan compared to the non-adaptive planned dosimetry
Impact of rectal spacers | Enrollment through 5 year follow up
  Physician reported toxicity and patient reported outcomes with or without implanted resorbable rectal spacer

OTHER OUTCOMES:
Decipher prognostic ability | 5 years after end of SBRT
  Correlation of the Decipher risk category (low/intermediate/high) with biochemical recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Leeman, MD, Principal Investigator — Brigham and Women's Hospital; Jeremy Bredfeldt, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (7):
- United States (5):
  - Duarte Cancer Center, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Universitätsklinikum des Saarlandes (Saarland Univerisity Hospital), Homburg, Saarland, Germany
- Hospital Universitario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No